CLINICAL TRIAL: NCT05048316
Title: Pilot Study to Develop a Group-Based E-Health Intervention for Young Adult Cancer Survivors
Brief Title: Study to Develop a Group-Based E-Health Intervention for YA Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MCC-21053
Record Dates: First submitted 2021-08-31; First posted 2021-09-17 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Cancer Survivor; Young Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- eHealth (Experimental): Weekly video conference groups led by a trained facilitator
  Interventions: Behavioral: Cognitive-Behavioral Stress Management and Health Education

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Stress Management and Health Education — Participants will attend group sessions with a trained facilitator held over videoconference. Sessions will each last 2 hours and will be held once weekly for 10 weeks. Sessions will include Cognitive-Behavioral Stress Management and health education content.

SUMMARY:
Investigators will test an evidence-based behavioral intervention that is responsive to Young Adults (YA's) expressed needs and priorities

ELIGIBILITY:
Inclusion Criteria:

* 18-39 years old
* Diagnosed with cancer between 18-39 years old
* Cancer diagnosis was non-metastatic
* Completed cancer treatment between 1 month and 5 years prior to enrollment, with the exception of ongoing hormone therapy
* No documented or observable psychiatric or neurological disorders that could interfere with participation (e.g., active psychosis, active substance abuse), as identified by the referring medical team, chart review, or screening
* Able to speak and read English
* Able to provide informed consent

Exclusion Criteria:

* Metastatic disease
* Continued cancer treatment
* Psychiatric or neurological disorders that could interfere with study participation
* Vulnerable populations will not be included

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2022-01-06 (Actual); Study Completion 2022-01-06 (Actual)

PRIMARY OUTCOMES:
Satisfaction assessed by study-specific survey during the intervention - Acceptability | During intervention
  The intervention will be deemed acceptable if, on average, participants report satisfaction with the weekly sessions as ≥2 on a 0-4 scale.
Satisfaction assessed by study-specific survey after the intervention - Acceptability | Immediately after the intervention
  The intervention will be deemed acceptable if, on average, participants report satisfaction with the overall program and intent to continue using the intervention skills as ≥2 on a 0-4 scale.
Session attendance after the intervention - Acceptability | Immediately after the intervention
  Videoconference delivery will be acceptable if average group attendance is ≥6/10 sessions.

SECONDARY OUTCOMES:
Quality of life before intervention | Baseline
  Participants will complete the 27-item Functional Assessment of Cancer Therapy - General
Change in quality of life at after intervention | Immediately after intervention
  Participants will complete the 27-item Functional Assessment of Cancer Therapy - General

OTHER OUTCOMES:
Symptom burden before intervention | Baseline
  Participants will complete the 22-item Impact of Event Scale-Revised
Change in Symptom burden after intervention | Immediately after intervention
  Participants will complete the 22-item Impact of Event Scale-Revised
Cancer-related distress before intervention | Baseline
  Participants will complete the 22-item Impact of Event Scale-Revised
Change in cancer-related distress after intervention | Immediately after intervention
  Participants will complete the 22-item Impact of Event Scale-Revised
Stress management skills self-efficacy before intervention | Baseline
  Participants will complete subscales from the Measure of Current Status
Change in stress management skills self-efficacy after intervention | Immediately after intervention
  Participants will complete subscales from the Measure of Current Status
Coping before intervention | Baseline
  Participants will complete the Brief-COPE
Change in coping after intervention | Immediately after intervention
  Participants will complete the Brief-COPE

CONTACTS AND LOCATIONS:
Overall Officials: Laura Oswald, PhD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fox RS, Badger TA, Moya S, Gudenkauf LM, Nelson MA, O'Neill RM, Leete JJ, Friedman SE, Katsanis E, Victorson DE, Sanford SD, Penedo FJ, Antoni MH, Oswald LB. An HRQOL Proof-Of-Concept Analysis of the eHealth TOGETHER Intervention for Adolescent and Young Adult Cancer Survivors: A Brief Report. Psychooncology. 2025 Jul;34(7):e70234. doi: 10.1002/pon.70234. PMID 40879639
- [Derived] Oswald LB, Lyleroehr M, Gudenkauf LM, Armstrong GE, Tometich DB, Sanford SD, Loecher N, Geiss C, Rodriguez Y, Scheel KL, Nieves-Lopez A, Jim HSL, Gonzalez BD, Antoni MH, Penedo FJ, Reed D, Katsanis E, Salsman JM, Victorson D, Fox RS. Development and initial testing of TOGETHER-YA: an eHealth-delivered and group-based psychosocial intervention for young adult cancer survivors. Support Care Cancer. 2022 Dec;30(12):10067-10076. doi: 10.1007/s00520-022-07382-y. Epub 2022 Oct 14. PMID 36229547
- See also: Moffitt Clinical Trial Search — https://moffitt.org/clinical-trials-research/clinical-trials/

DOCUMENTS (1):
  • Informed Consent Form (2021-08-25): https://cdn.clinicaltrials.gov/large-docs/16/NCT05048316/ICF_000.pdf